CLINICAL TRIAL: NCT05525156
Title: The Effect of Aspirin on HIV Disease Progression Among HIV- Infected Individuals Initiating Anti- Retroviral Therapy
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The study stopped due to expiry of study drugs
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); Kumamoto University (Other)
Responsible Party: Principal Investigator, Tosi Michael Mwakyandile, Principal Investigator, Muhimbili University of Health and Allied Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DA.282/298/01 /C; PACTR202003522049711 (Registry Identifier: Pan African Clinical Trial Registry); R25TW011227 (NIH); 5D43TW009775-03 (NIH)
Record Dates: First submitted 2022-08-28; First posted 2022-09-01 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Hiv; Cardiovascular Diseases
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin arm (Experimental): In addition to their antiretroviral regimen, participants self administer blister packaged enteric coated tablet of 75 mg aspirin (Cardisprin 75, Cosmos, Nairobi, Kenya) for 24 weeks at a dose of one tablet per day at evening times swallowed wholly with a glass of clean drinking water, preferably after a meal. All adults initiating antiretroviral therapy are prescribed the default combination of tenofovir (TDF) +lamivudine (3TC)+dolutegravir (DTG). Those with contraindications are alternatively prescribed abacavir+3TC+DTG or TDF +3TC+efavirenz and in special situations zidovudine+3TC+DTG
  Interventions: Drug: aspirin enteric coated tablet 75 mg
- Placebo arm (Placebo Comparator): In addition to their antiretroviral regimen, participants self administer blister packaged placebo (Cardisprin 75, Cosmos, Nairobi, Kenya) for 24 weeks at a dose of one tablet per day at evening times swallowed wholly with a glass of clean drinking water, preferably after a meal. The placebo has colour, shape and size similar to aspirin
  Interventions: Drug: aspirin enteric coated tablet 75 mg

INTERVENTIONS:
Drug: aspirin enteric coated tablet 75 mg — blister packaged enteric coated tablet of 75 mg aspirin taken once daily for 24 weeks in addition to the conventional antiretroviral drugs
  Other Names: antiretroviral drugs

SUMMARY:
Introduction An increase in cardiovascular disease (CVD) among people living with HIV infection is linked to platelet and immune activation, a phenomenon unabolished by antiretroviral (ARV) drugs alone. In small studies, aspirin (acetylsalicylic acid [ASA]) has been shown to control immune activation, increase CD4+ count, halt HIV disease progression and reduce HIV viral load (HVL). The investigators present a protocol for a larger suspended randomised placebo controlled trial on the effect of an addition of ASA to ARV drugs on HIV disease progression.

Methods and analysis A single-centre phase IIA double-blind, parallel-group randomised controlled trial intended to recruit 454 consenting ARV drug-naïve, HIV-infected adults initiating ART. Participants were randomised in blocks of 10 in a 1:1 ratio to receive, in addition to ARV drugs, 75 mg ASA or placebo for 6 months. The primary outcome is the proportion of participants attaining HVL of <50 copies/mL by 8, 12 and 24 weeks. Secondary outcomes include proportions of participants with HVL of >1000 copies/mL at week 24, attaining a >30% rise of CD4 count from baseline value at week 12, experiencing adverse events, with normal levels of biomarkers of platelet and immune activation at weeks 12 and 24 and rates of morbidity and all-cause mortality. Intention-to-treat analysis will be done for all study outcomes.

DETAILED DESCRIPTION:
Despite the introduction of antiretroviral (ARV) therapy, HIV is still a public health problem in Eastern and Southern Africa. The wide spread use of the ARV drugs has improved the life expectancy of people living with HIV and/ or acquired immunodeficiency syndrome (AIDS). As a result, there has been an increase in the prevalence of and mortality from non - AIDS complications such as non - AIDS defining cancers, liver, pulmonary and cardiovascular diseases. The increase in the non - AIDS complications especially the cardiovascular disease risk is linked to platelet and immune activation. Antiretroviral therapy (ART) does not completely abolish the immune activation and the platelet activation making it a necessity to find additional therapy to the conventional ART therapy, that will decrease the occurrence of these non- AIDS complications and their associated morbidities. Aspirin or acetyl salicylic acid (ASA) has shown promise as such an additional drug. In addition, ASA appears to have an array of beneficial effects in the HIV infected individuals. ASA is reported to possibly cause a reduction in HIV load, increase CD4 counts and halt the clinical HIV disease progression. Literature shows that additional therapy to ARV drugs may compromise adherence to ART among HIV- infected individuals. However, when addition of a pill is associated with significant benefit, the addition of a pill or pills may be justifiable. For example, addition of medication for opportunistic infection, methadone maintenance therapy and antidepressants has been reported to improve adherence to ART among HIV- infected patients in some studies. Therefore, considering the reported benefits of ASA in the HIV- infected population, it is important to study the effect of the addition of ASA on both the HIV disease progression and the adherence to ARV drugs. The project aims at investigating the effects of low dose aspirin on immunological, virologic and clinical outcomes among HIV- infected individuals initiating ART.

The investigators hypothesize that addition of ASA to ART in the newly recruited HIV- infected patients will be associated with earlier and sustained virologic suppression, better immunological and clinical responses and improved quality of life. And also that addition of ASA to ART in the newly recruited HIV- infected patients will not compromise adherence to ARV therapy.

b. The objectives of the research project: Broad objective: To determine the effect of low dose of ASA on HIV disease progression and adherence to anti- retroviral therapy among HIV-infected individuals initiating ARV therapy.

Specific Objectives i. To compare the HIV viral loads measured at 2, 3 and 6 months among HIV- infected individuals after initiating ARV therapy alone or ARV therapy and 75mg ASA.

ii. To compare the CD4 counts measured at 3 and 6 months among HIV- infected individuals after initiating ARV therapy alone or ARV therapy and 75mg ASA.

iii. To compare the plasma levels of immune activation biomarker (sCD14) measured at 3 and 6 months among HIV- infected individuals after initiating ARV therapy alone or ARV therapy and 75mg ASA.

iv. To compare the plasma levels of platelet activation biomarker (P- selectin) measured at 3 and 6 months among HIV- infected individuals after initiating ARV therapy alone or ARV therapy and 75mg ASA.

v. To compare percentage of activated T cells (CD38 positive and HLA-DR positive T cells) measured at 3 and 6 months among HIV- infected individuals after initiating ARV therapy alone or ARV therapy and 75mg ASA.

vi. To compare percentages of exhausted T cells (PD1 positive T cells) measured at 3 and 6 months among HIV- infected individuals after initiating ARV therapy alone or ARV therapy and 75mg ASA.

vii. To compare morbidity among HIV- infected individuals initiating ARV therapy alone or ARV therapy and 75mg ASA.

viii. To compare all-cause-mortality among HIV- infected individuals initiating ARV therapy alone or ARV therapy and 75mg ASA.

ix. To determine level of adherence to ARV therapy among HIV- infected individuals initiating ARV therapy and ASA or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Consenting newly recruited male or female HIV-infected patients
* Antiretroviral drug-naïve initiating on antiretroviral drugs
* Age 18 years or older
* Willingness to stay in Dar es Salaam for at least 6 consecutive months
* Willingness to attend HIV clinics at Temeke or Mbagala Rangi Tatu or Mwananyamala hospital for at least six consecutive months

Exclusion Criteria:

* Previous intolerance or allergy to aspirin or any aspirin products
* Asthmatics
* Predisposition to bleeding (increased chance of bleeding due to being on antiplatelets and/or anticoagulants and/or having history of or active diagnosis of bleeding disorder)
* Antithrombotic therapy
* Therapy with protocol prohibited drugs
* Active or history of peptic ulcer disease
* Pregnancy
* Severe renal disease (eGFR <30 mil/min/1.73 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 454 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-06-22 (Estimated)

PRIMARY OUTCOMES:
Virologic suppression | 8 weeks
  The primary outcome is the proportion of participants attaining viral load of <50 copies/mL at the end of 8, 12 and 24 weeks. I

SECONDARY OUTCOMES:
Virologic failure, safety, immunological and clinical responses | up to 24 weeks for safety, 12 and 24 weeks
  Secondary outcomes include proportion of participants with viral load of >1000 copies/mL at the end of 24 weeks, proportion of participants attaining a >30% rise of CD4 count from baseline value at the end of 12 weeks, and prevalence of morbidity and all-cause mortality. Other secondary outcomes are proportion of participants with normal levels of the assessed biomarkers of platelet and immune activation at the end of 12 and 24 weeks, proportion of participants experiencing adverse events, mean percentage adherence to antiretroviral drugs and mean percentage compliance to the study drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Eligius F Lyamuya, MD, MMed, PhD, FTAAS, FCPath, Principal Investigator — Muhimbili University of Health and Allied Sciences
Locations (1):
- Mwananyamala Regional Referral Hospital, Mbagala Rangi Tatu Hospital, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the respective article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From 9 months and to 36 months after article publication
Access Criteria: Investigators with approval by an independent review committee for proposed use of data. Data will be shared for individual participant data meta analysis The mechanism by which data will be made available is that proposals may be submitted up to 36 months after respective article publication. after this period data will be made available at MUHAS data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Mwakyandile T, Shayo G, Mugusi S, Sunguya B, Sasi P, Moshiro C, Mugusi F, Lyamuya E. Effect of aspirin on HIV disease progression among HIV-infected individuals initiating antiretroviral therapy: study protocol for a randomised controlled trial. BMJ Open. 2021 Nov 2;11(11):e049330. doi: 10.1136/bmjopen-2021-049330. PMID 34728445
- [Derived] Mwakyandile TM, Shayo GA, Sasi PG, Kunambi PP, Mugusi FM, Barabona G, Ueno T, Lyamuya EF. Low-dose aspirin is not effective as an adjunct treatment for HIV infection among people living with HIV on dolutegravir-based antiretroviral therapy: A randomised double-blind, parallel-group placebo-controlled trial. PLoS One. 2025 Aug 29;20(8):e0331087. doi: 10.1371/journal.pone.0331087. eCollection 2025. PMID 40880360
- See also: study protocol paper — http://bmjopen.bmj.com/cgi/content/full/bmjopen-2021-049330